CLINICAL TRIAL: NCT01125956
Title: Improving Diabetes Control Through Peer Counseling and Incentives
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01164
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes; Diabetes mellitus; HbA1c
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): This group will receive usual diabetes care through their primary care clinicians.
- Peer counseling (Experimental): A peer counselor will be assigned to each participant who currently has good diabetes control but had poor control in the past 3 years.
  Interventions: Behavioral: Assigned a peer counselor
- Financial incentives (Experimental): Patient participants in the financial incentive arm will be given $100 for reduction of HbA1c by 1 point in a 6 month period and $200 for reduction by 2 points.
  Interventions: Behavioral: Financial incentives

INTERVENTIONS:
Behavioral: Assigned a peer counselor — Dyads will be given $20 per month if they have contact 4 or more times during a month.
  Arms: Peer counseling
Behavioral: Financial incentives — Participants will be given $100 for reduction of HbA1c by 1 point in a 6 month period and $200 for reduction by 2 points.
  Arms: Financial incentives

SUMMARY:
The specific aims of this study are to test whether in a cohort of low-income minority veterans with poor diabetes mellitus (DM) control:

1. Peer counseling is an effective means of reducing HbA1c (a measure of glucose control).
2. Financial incentives are an effective means of reducing HbA1c. This is a randomized controlled pilot study. There will be 3 arms: 1) a control group of poorly controlled diabetics getting usual care; 2) peer counseling with no incentives; and 3) financial incentives without peers. Ultimately, contingent on the success of this intervention, the researchers plan to apply for funding for a large scale intervention employing both peer counseling and incentives to improve DM control in low income and minority patients who are at high risk for premature morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* African American veteran
* 50-70 years old
* ICD-9CM diagnosis code consistent with DM (any ICD-9CM code starting with 250)
* For patients: last two HbA1c greater than 8% with at least one measure being within 3 months of enrollment
* For peer counselors: HbA1c of greater than 8% in the past 3 years and an HbA1c less than or equal to 7.5% within 3 months of enrollment

Exclusion Criteria:

* Unstable medical condition that would likely prevent the subject from completing the study
* Patients enrolled in Telehealth will be excluded as such enrollment does not constitute usual care

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | Baseline, 6 months
  Change in HbA1c from baseline will be the primary outcome measure.

SECONDARY OUTCOMES:
Counts of the number of hypoglycemic events | 6 months
  All events and serious events related to hypoglycemia will be counted over the 6 month intervention period, including emergency room visits and hospitalizations.
Number of peer encounters | 6 months
  The number of peer encounters by arm will be described.
Experience of peer counseling | 6 months
  The experience of peer counseling from both poorly controlled diabetics and counselors will be described.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Long, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Philadelphia Veterans Affairs Medical Center, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Long JA, Jahnle EC, Richardson DM, Loewenstein G, Volpp KG. Peer mentoring and financial incentives to improve glucose control in African American veterans: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):416-24. doi: 10.7326/0003-4819-156-6-201203200-00004. PMID 22431674
- See also: LDI Center for Health Incentives — http://www.med.upenn.edu/ldichi/
- See also: VA Center for Health Equity and Promotion (CHERP) — https://www.cherp.research.va.gov/
- See also: This research was supported by a grant from the National Institute on Aging, P30-AG036592. The content is solely the responsibility of the authors and does not necessarily represent the official views of the National Institute on Aging or the NIH — https://grants.nih.gov/grants/guide/rfa-files/RFA-AG-09-005.html